CLINICAL TRIAL: NCT01600586
Title: A Pacifier-Activated Music Player With Mother's Voice Improves Oral Feeding in Preterm Infants
Brief Title: A Clinical Trial of A Pacifier-Activated Music Player
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Vanderbilt Kennedy Center (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VKC 4-30-100-9622; UL1RR024975-01 (NIH)
Record Dates: First submitted 2012-05-09; First posted 2012-05-17 (Estimated); Results first posted 2018-05-07 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Prematurity
Keywords: Neonatal Intensive Care Unit (NICU); Music therapy; Premature infant; Oral feeds; Non-Nutritive Sucking; Suck rate; Suck efficiency; Contingent music; Mother's voice
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pacifier-Activated-Lullaby system (PAL) (Experimental): Pacifier-Activated-Lullaby system (PAL) group.
  Interventions: Device: Pacifier-Activated-Lullaby system (PAL).
- No PAL group (No Intervention): No PAL. Standard of care procedures.

INTERVENTIONS:
Device: Pacifier-Activated-Lullaby system (PAL). — Pacifier-Activated-Lullaby system (PAL).
  Arms: Pacifier-Activated-Lullaby system (PAL)

SUMMARY:
Neonatal intensive care unit infants are at high risk for oromotor difficulties including poor coordination of sucking swallowing and breathing. These feeding difficulties often result in prolonged hospitalization, with increased physiologic stressors and poor growth. In preliminary studies, Pacifier Activated Lullaby (PAL) use showed potential increased oromotor skills and decreased length of hospitalization.

The investigators propose to test the hypothesis that a week-long PAL intervention can improve feeding skills and decrease stress compared to standard of care parental interactions in infants in the late preterm period. The investigators also hypothesize that these improvements will result in shorter hospital stays and increased growth in the intervention group.

Our study design is a prospective randomized controlled trial design of 94 infants (Post-conceptional ages 34-36 weeks). The 47 intervention-group infant/mother dads will receive a book library with one lullaby book and record her voice to the PAL, which the music therapist will then administer in 15-minute sessions for 5 consecutive days. The 47 participants in the control group will receive the same library but no recording will be made or PAL used. Outcomes measured will include time to full oral feeds, suck rate and efficiency, salivary cortisol levels before and after intervention, daily growth parameters and nutritional data, and hospital length of stay.

DETAILED DESCRIPTION:
Objectives: We conducted a randomized trial to test the hypothesis that the mother's voice played through a pacifier-activated music (PAM) player during nonnutritive sucking would improve the development of sucking ability and promote more effective oral feeding in preterm infants.

Methods: Preterm infants between 34 0/7 and 35 6/7 weeks postmenstrual age, including those with brain injury, who were taking at least half their feedings enterally and less than half orally, were randomly assigned to receive 5 daily 15-minute sessions of either PAM with mother's recorded voice or no PAM, along with routine nonnutritive sucking and maternal care in both groups. Assignment was masked to the clinical team.

ELIGIBILITY:
Inclusion Criteria:

* All infants at 34 0/7 to 35 6/7 weeks post-conceptional age cared for in the Vanderbilt NICU who are receiving more than 50 % of their nutrition as enteral feeds, and are in individual rooms or in the room with their sibling.

Exclusion Criteria:

* infants on ventilators or Continuous Positive Airway Pressure (CPAP),
* infants determined to be unsafe to feed orally by the medical team or the feeding/speech specialists at Vanderbilt.

Ages: 34 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olena D Chorna, MM, MT-BC, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: PI has left Vanderbilt, data obtained from publication http://pediatrics.aappublications.org/content/133/3/462.full
Groups:
- Books, PAL Group: PAL group
  Pacifier-Activated-Lullaby system (PAL).: Pacifier-Activated-Lullaby system (PAL).
- Books, No PAL Group: No PAL
  At enrollment, all mother-infant dyads received a set of 4 well-known children's books, 2 of which were single-story songbooks. Mothers in both groups were encouraged to read and sing to their infants whenever they were present; no time quota, schedule, or log was provided. Mothers were informed that the study's objective was to evaluate the influence of their voice on their infant's feeding ability.
Period: Overall Study
Arm/Group | Books, PAL Group | Books, No PAL Group
Started | 49 | 51
Completed | 46 | 48
Not Completed | 3 | 3
Not completed — Physician Decision | 3 | 3

BASELINE CHARACTERISTICS:
Population: NICU infants
Groups:
- Books, PAL Group: PAL group
  Pacifier-Activated-Lullaby system (PAL).: Pacifier-Activated-Lullaby system (PAL).
  Infants were randomly assigned by using a block system to control or intervention groups. Eligible siblings were enrolled into the same group because they shared the same room in the NICU. If 1 child received the PAM intervention while the other engaged in NNS, diffusion of treatment might occur; removal of the siblings' pacifier during the pacifier-activated lullaby (PAL) was not an alternative acceptable to nursing staff.
- Books, No PAL Group: No PAL
- Total: Total of all reporting groups
Arm/Group | Books, PAL Group | Books, No PAL Group | Total
Number analyzed (Participants) | 46 | 48 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 46 | 48 | 94
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 25 | 47
  Male | 24 | 23 | 47
Region of Enrollment [Number; unit: participants]
  United States | 46 | 48 | 94
Birth weight, g, median [Median (Inter-Quartile Range); unit: grams] | 1495 [1122 to 1742] | 1405 [1057 to 1684] | 1450 [1100 to 1712]
White matter injury [Number; unit: number of participants] — White matter injury information was derived from the medical record, as approved by the Ethics board.
  number of participants | 7 | 9 | 16
Feeding rate at study start [Mean (Inter-Quartile Range); unit: ml/min] | 0.6 [0.4 to 0.8] | 0.6 [0.1 to 0.8] | 0.6 [0.25 to 0.8]
No. of oral feedings/d at study start [Median (Full Range); unit: feedings per day] | 2 [1 to 8] | 2 [1 to 8] | 2 [1 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Suck Rate and Efficiency: Change From Pre-test (Day 0) to Post-test (Day 5)
Description: Feeding rate when nippling was calculated by dividing the number of cc of nippled nutrition by time for consumption. This data was recorded at two time points: pre and post intervention
Time Frame: Day 0, and Day 5
Measure: Mean (Inter-Quartile Range); unit: mL/min
Groups:
- PAL Intervention: This group of participants received PAL intervention
- No PAL Intervention: This group of participants did not receive PAL intervention
Arm/Group | PAL Intervention | No PAL Intervention
Number analyzed (Participants) | 47 | 48
mL/min | 2.0 [1.5 to 2.3] | 0.9 [0.5 to 1.2]

2. Secondary Outcome: Discharge Weight
Description: Description: Growth measures.
Time Frame: day of hospital discharge (approximately 5-7 weeks)
Measure: Median (Inter-Quartile Range); unit: grams
Groups:
- This is the PAL Intervention: This group received intervention
- No PAL: This group received no PAL intervention
Arm/Group | This is the PAL Intervention | No PAL
Number analyzed (Participants) | 46 | 48
grams | 2000 [1892 to 2228] | 1990 [1902 to 2120]

3. Secondary Outcome: Change From Pre-test(Day 0)in Salivary Cortisol Levels to Post-test (Day 5)
Description: Description: Stress: Salivary cortisol levels at baseline and after 1 week of PAL in the intervention group.
Time Frame: Day 0, and Day 5
Population: Specific data is no longer available, Outcome is described here: http://pediatrics.aappublications.org/content/133/3/462.full
Groups:
- This is the PAL Intervention Group: This is the PAL intervention group
- This is the NO PAL Group: This is the NO PAL group
Arm/Group | This is the PAL Intervention Group | This is the NO PAL Group
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Hospital Length of Stay
Description: Description: Data on hospital stay was recorded from the chart. The participants were be followed for the duration of the hospital stay from the time of consent for participation to the time discharge from the NICU is documented.
Time Frame: days from consent to discharge
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Books, PAL Group | Books, No PAL Group
Number analyzed (Participants) | 46 | 48
days | 41 [25 to 69] | 50 [31 to 86]

5. Secondary Outcome: Number of Days to Full Oral Feeds
Description: Aim: Quantify the effect of the PAL intervention on efficiency of sucking and time to reaching full oral feeds in comparison to controls. Data on the number of days from Day 0 of the study to the date of first documented full oral feed, up to 70 days (or date of death from any cause) were be recorded from the chart.
Time Frame: Day 0 of the study to the date of first documented full oral feed (up to 70 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Books, PAL Group | Books, No PAL Group
Number analyzed (Participants) | 46 | 48
days | 31 [17 to 54] | 38 [24 to 69]

ADVERSE EVENTS:
Groups:
- PAL Group: PAL group
  Pacifier-Activated-Lullaby system (PAL).: Pacifier-Activated-Lullaby system (PAL).
Arm/Group | PAL Group | Books, No PAL Group
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/48
Other Adverse Events (participants affected / at risk) | 0/46 | 0/48

LIMITATIONS AND CAVEATS:
PI left Vanderbilt, data obtained from publication http://pediatrics.aappublications.org/content/133/3/462.full

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No